CLINICAL TRIAL: NCT00055445
Title: IdB 1016 in Hepatitis C
Brief Title: IdB 1016 Treatment for Hepatitis C Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000992-01A1 (NIH); IdB-1016-UW-001
Record Dates: First submitted 2003-03-03; First posted 2003-03-04 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Hepatitis C, Chronic
Keywords: Complementary Therapies; IdB 1016; Silybin; Antioxidant; Hepatitis C Virus; Phosphatidylcholine
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — IdB 1016

INTERVENTIONS:
Drug: IdB 1016

SUMMARY:
This study will measure the safety and tolerability of three different doses of IdB 1016 in patients with hepatitis C disease who have not responded to or are poor candidates for interferon-based therapies.

NOTE: THE STUDY WILL ONLY RECRUIT STUDY PARTICIPANTS AT UNIVERSITY OF WASHINGTON MEDICAL CENTER IN SEATTLE

DETAILED DESCRIPTION:
Results from two open label and four randomized placebo-controlled studies in patients with liver disease of diverse etiology suggest that IdB 1016 (oral silybin-phosphatidylcholine phytosome) is well tolerated and significantly improves serum liver enzyme levels. However, IdB 1016 dosing in these studies ranged from 314 mg bid to 314 mg tid, which is below Phase I doses that were well tolerated in healthy volunteers. None of the studies tested the safety and efficacy of IdB 1016 strictly in patients with chronic hepatitis C disease or measured post-treatment histologic changes.

This study will be an open label, randomized, dose-finding study. There will be three arms corresponding to three different IdB 1016 doses: 314 mg, 624 mg, and 942 mg tid. Each arm will have 15 patients diagnosed with chronic hepatitis C and will be stratified to five patients with fibrosis stage II (periportal fibrosis), five patients with fibrosis stage III (bridging fibrosis), and five patients with fibrosis stage IV (compensated cirrhosis). The treatment duration will be 12 weeks. Patients will be followed for an additional 4 weeks after treatment cessation to assess residual effects of measured parameters. Patients will have clinic visits on Day -21 (screening), Day 1 (treatment initiation), Day 29, Day 57, Day 85 (end of treatment), and Day 113 (follow-up after washout).

ELIGIBILITY:
Inclusion Criteria:

* HCV infection according to ELISA-2
* Detectable HCV RNA PCR as measured within the previous 6 months
* Poor responders to, inadequate candidates for, or unwilling to use interferon-based therapies
* Serum ALT >= 1.3 times above normal
* Persistently elevated serum ALT levels according to two measures in the previous 12 months
* Evidence of stage II (periportal fibrosis), III (bridging fibrosis), or IV (compensated cirrhosis) in the Batts-Ludwig scoring system according to a liver biopsy performed in the last 2 (stage II and III patients) to 5 (stage IV patients) years. Patients with clinical signs of compensated cirrhosis (portal hypertension, non-bleeding varices) do not require a biopsy.
* Able and willing to follow protocol directions for the duration of the study
* Able and willing to maintain a consistent lifestyle routine (e.g., diet, exercise, medications, and dietary supplements) and sleep schedule for the duration of the study
* Able and willing to stop taking dietary supplements outside the study protocol for the duration of the study
* Able and willing to practice two methods of contraception during the study period, including the 4 week follow-up. This applies to women with childbearing potential and men whose sexual partners have childbearing potential.

Exclusion Criteria:

* Pregnant or breastfeeding
* Liver synthetic dysfunction (albumin < 3.2 g/dL, total bilirubin > 3.0 mg/dL, prothrombin time > 1.5 seconds prolonged)
* History of ascites, variceal bleeding, encephalopathy, jaundice, or extrahepatic biliary obstruction
* History of uncontrolled diabetes mellitus
* Known concomitant acute or chronic viral liver infections (e.g., hepatitis A, hepatitis B, Epstein-Barr, or cytomegalovirus)
* Concomitant autoimmune and inflammatory disease (e.g., rheumatoid arthritis, lupus)
* Other types of concomitant liver disease
* HIV-1 coinfection
* Chronic use of hepatotoxic drugs (e.g., acetaminophen)
* Interferon-based therapies in the past 6 months
* Alcohol consumption within 3 months prior to entry. Patients with a history of alcohol abuse should be at least 2 years into recovery.
* Use of recreational oral or IV drugs. Patients with a history of drug addiction should be at least 2 years into recovery.
* History of untreated malignancy
* Remission from previous malignant neoplasms <= 6 months
* History of significant renal, endocrine, cardiac, or pulmonary disease
* Use of supplements containing compounds derived from milk thistle
* Proven allergy to milk thistle or any derived compounds
* Subjects taking warfarin or coumadin due to silybin's potential interactions with cytochrome CYP 29C
* Any condition or concomitant medication or supplement that could hinder the outcomes of the study or the safety of the patient as determined by the principal investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2003-11; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Kris V. Kowdley, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Carini R, Comoglio A, Albano E, Poli G. Lipid peroxidation and irreversible damage in the rat hepatocyte model. Protection by the silybin-phospholipid complex IdB 1016. Biochem Pharmacol. 1992 May 28;43(10):2111-5. doi: 10.1016/0006-2952(92)90168-i. PMID 1599497
- [Background] Comoglio A, Tomasi A, Malandrino S, Poli G, Albano E. Scavenging effect of silipide, a new silybin-phospholipid complex, on ethanol-derived free radicals. Biochem Pharmacol. 1995 Oct 12;50(8):1313-6. doi: 10.1016/0006-2952(95)02001-s. PMID 7488251
- [Background] Conti M, Malandrino S, Magistretti MJ. Protective activity of silipide on liver damage in rodents. Jpn J Pharmacol. 1992 Dec;60(4):315-21. doi: 10.1254/jjp.60.315. PMID 1287266
- [Background] Edwards J, Grange LL, Wang M, Reyes E. Fetoprotectivity of the flavanolignan compound siliphos against ethanol-induced toxicity. Phytother Res. 2000 Nov;14(7):517-21. doi: 10.1002/1099-1573(200011)14:73.0.co;2-w. PMID 11054841
- [Background] Morazzoni P, Montalbetti A, Malandrino S, Pifferi G. Comparative pharmacokinetics of silipide and silymarin in rats. Eur J Drug Metab Pharmacokinet. 1993 Jul-Sep;18(3):289-97. doi: 10.1007/BF03188811. PMID 8149949
- [Background] Morazzoni P, Magistretti MJ, Giachetti C, Zanolo G. Comparative bioavailability of Silipide, a new flavanolignan complex, in rats. Eur J Drug Metab Pharmacokinet. 1992 Jan-Mar;17(1):39-44. doi: 10.1007/BF03189986. PMID 1499596
- [Background] Comoglio A, Leonarduzzi G, Carini R, Busolin D, Basaga H, Albano E, Tomasi A, Poli G, Morazzoni P, Magistretti MJ. Studies on the antioxidant and free radical scavenging properties of IdB 1016 a new flavanolignan complex. Free Radic Res Commun. 1990;11(1-3):109-15. doi: 10.3109/10715769009109673. PMID 2074043
- [Background] Barzaghi N, Crema F, Gatti G, Pifferi G, Perucca E. Pharmacokinetic studies on IdB 1016, a silybin- phosphatidylcholine complex, in healthy human subjects. Eur J Drug Metab Pharmacokinet. 1990 Oct-Dec;15(4):333-8. doi: 10.1007/BF03190223. PMID 2088770
- [Background] Schandalik R, Perucca E. Pharmacokinetics of silybin following oral administration of silipide in patients with extrahepatic biliary obstruction. Drugs Exp Clin Res. 1994;20(1):37-42. PMID 7924893
- [Background] Schandalik R, Gatti G, Perucca E. Pharmacokinetics of silybin in bile following administration of silipide and silymarin in cholecystectomy patients. Arzneimittelforschung. 1992 Jul;42(7):964-8. PMID 1329780
- [Background] Buzzelli G, Moscarella S, Giusti A, Duchini A, Marena C, Lampertico M. A pilot study on the liver protective effect of silybin-phosphatidylcholine complex (IdB1016) in chronic active hepatitis. Int J Clin Pharmacol Ther Toxicol. 1993 Sep;31(9):456-60. PMID 8225695